CLINICAL TRIAL: NCT03422003
Title: Study of Radiation Fractionation on Patient Outcomes After Breast REConstruction (FABREC) for Invasive Breast Carcinoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Rinaa Punglia, MD, MPH, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-304
Record Dates: First submitted 2018-01-19; First posted 2018-02-05 (Actual); Results first posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Radiation; Hypofractionation; Randomization
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm 1: Hypofractionation (Experimental): 16 fractions of radiation therapy (daily, Monday through Friday) to the chest wall with or without internal mammary nodes, and 15 fractions to the supraclavicular (with or without axillary) lymph nodes.
  Interventions: Radiation: Radiation Therapy
- Arm 2: Conventional Radiation Therapy (Active Comparator): 25 fractions of radiation therapy (daily, Monday through Friday) to the chest wall with or without internal mammary nodes, and 23-25 fractions to the supraclavicular (with or without axillary) lymph nodes.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — For the conventional fractionation arm: Each fraction will consist of 200 cGy per day. Total dose = 5000 cGy to the chest wall and 4600-5000 cGy to the lymph nodes.
  For the hypofractionation arm: Each fraction consists of 266 cGy per day. Total dose = 4256 cGy to the chest wall and 3990 cGy to the lymph nodes.

SUMMARY:
This study is a randomized trial of hypofractionation (short-course) radiation therapy versus conventional radiation therapy in women who have undergone mastectomy and immediate breast reconstruction. The investigators will assess cosmetic and reconstruction outcomes, lymphedema, cancer status, side effects, and oncologic outcomes.

DETAILED DESCRIPTION:
Over 180,000 diagnoses of invasive breast cancer are made in the US each year. Over one-third of women with early stage and over half with late-stage breast cancer are treated with mastectomy (removal of the entire breast) due to tumor size, multiple cancers within the breast, genetic cancer predisposition, and/or patient preference. Following treatment with mastectomy, women who receive breast reconstructive surgery may experience better quality of life as they do not have to leave surgery with a bare chest wall. However, large randomized trials of post-mastectomy radiation therapy reveal a survival benefit with the addition of radiation after mastectomy in women who have cancer present in the axillary lymph nodes (6). The delivery of radiation therapy in the presence of a breast reconstruction is challenging and often leads to undesirable consequences including reconstruction loss, need for major surgical revision, or poor cosmetic outcomes. Therefore, oncologists and patients are forced to decide between the potential for improved oncologic outcomes with radiation therapy versus increased likelihood of complications and suboptimal cosmetic results. Because of this, some patients may be foregoing reconstruction if radiation therapy after mastectomy is needed; or foregoing radiation therapy if they have had breast reconstructive surgery (28).

Hypofractionation enhances patient convenience and decreases treatment burden. This regimen has been shown in randomized trials largely in the breast-conservation setting to reduce acute radiation therapy side-effects, decrease fatigue at six months and improve cosmetic results (21, 22). Despite these results, adoption of hypofractionation has been slow among women with breast cancer treated with breast-conserving surgery (24, 25) likely due to familiarity and experience of conventional long-course radiation therapy.

While hypofractionation is used commonly in the UK for patients with mastectomy, there are no randomized studies particularly studying outcomes following shorter course radiation therapy in women who undergo mastectomy with breast reconstruction. Therefore, there is an even greater barrier to the use of hypofractionation in this setting in the US. With improved cosmetic results found with hypofractionation, this shorter regimen may have the potential to improve reconstruction success rates which are unfortunately modest overall, for patients who require post-mastectomy radiation. Especially in contrast to financial disincentives to reduce number of radiation treatments, Level I randomized evidence is needed in this population to change practice patterns regarding radiation regimen.

Our study of radiation fractionation regimens has the potential to increase use of hypofractionation among women treated with mastectomy, thereby decreasing treatment burden. Our team of patient stakeholders ensures that our outcomes measures encompass all domains of survivorship after breast cancer (physical and mental health as well as satisfaction with the decision-making process). Despite the large numbers of breast cancer survivors who undergo mastectomy, reconstruction and radiation therapy, little is known about which domains of quality of life are affected and their importance to these patients. This study uses previously validated tools for measuring patient outcomes, and have added questions for areas which are important to patients that may not have been captured adequately by previous tools. In concert with the increasing awareness of the importance of survivorship care to cancer care, identifying a comprehensive set of outcomes measurement tools following treatment with radiation therapy, mastectomy, and reconstruction is an important asset for future treatment evaluation in these women.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with clinical or pathologic stage I-III invasive breast cancer with TX-T3 tumor
2. Has been treated with mastectomy
3. Has undergone immediate reconstructive surgery with placement of a tissue expander or permanent implant at time of mastectomy
4. Is a candidate for unilateral post-mastectomy radiation therapy as per National Comprehensive Cancer Network (NCCN) guidelines (post-mastectomy radiation therapy is indicated for most patients with positive lymph nodes at time of surgery and infrequently for selected node-negative patients)
5. Use of bolus is permitted, but not required
6. Age ≥18

Exclusion Criteria:

1. T4 cancer
2. Recurrent breast cancer or history of prior breast radiation therapy
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, and/or mental health illness that the consenting investigator feels would affect patient's ability to participate in this study
4. Pregnant or nursing
5. History of a different malignancy except for the following circumstances:

   * Disease-free for at least five years and deemed by the investigator to be at low risk for recurrence of that malignancy (<5 %).
   * Cervical cancer in situ and basal cell or squamous cell carcinoma of the skin
6. Breast cancer requiring bilateral breast/chest wall radiation therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2030-04-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rinaa Punglia, MD MPH, Study Chair — Dana-Farber Cancer Institute; Julia Wong, MD, Study Chair — Dana-Farber Cancer Institute
Locations (15):
- United States (15):
  - University of California, San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Vail Health, Edwards, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Johns Hopkins Medicine, Washington D.C., District of Columbia
  - Eastern Maine Medical Center, Brewer, Maine
  - Maine Medical Center, Scarborough, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital/North Shore Center for Outpatient Care, Danvers, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center (DF/BWCC) at Milford Regional Medical Center, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center in clinical affiliation with South Shore Hospital, South Weymouth, Massachusetts
  - Lifespan/Rhode Island Hospital, Providence, Rhode Island
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] EBCTCG (Early Breast Cancer Trialists' Collaborative Group); McGale P, Taylor C, Correa C, Cutter D, Duane F, Ewertz M, Gray R, Mannu G, Peto R, Whelan T, Wang Y, Wang Z, Darby S. Effect of radiotherapy after mastectomy and axillary surgery on 10-year recurrence and 20-year breast cancer mortality: meta-analysis of individual patient data for 8135 women in 22 randomised trials. Lancet. 2014 Jun 21;383(9935):2127-35. doi: 10.1016/S0140-6736(14)60488-8. Epub 2014 Mar 19. PMID 24656685
- [Background] Duxbury PJ, Gandhi A, Kirwan CC, Jain Y, Harvey JR. Current attitudes to breast reconstruction surgery for women at risk of post-mastectomy radiotherapy: A survey of UK breast surgeons. Breast. 2015 Aug;24(4):502-12. doi: 10.1016/j.breast.2015.05.002. Epub 2015 May 26. PMID 26021276
- [Background] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial A of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet Oncol. 2008 Apr;9(4):331-41. doi: 10.1016/S1470-2045(08)70077-9. Epub 2008 Mar 19. PMID 18356109
- [Background] Shaitelman SF, Schlembach PJ, Arzu I, Ballo M, Bloom ES, Buchholz D, Chronowski GM, Dvorak T, Grade E, Hoffman KE, Kelly P, Ludwig M, Perkins GH, Reed V, Shah S, Stauder MC, Strom EA, Tereffe W, Woodward WA, Ensor J, Baumann D, Thompson AM, Amaya D, Davis T, Guerra W, Hamblin L, Hortobagyi G, Hunt KK, Buchholz TA, Smith BD. Acute and Short-term Toxic Effects of Conventionally Fractionated vs Hypofractionated Whole-Breast Irradiation: A Randomized Clinical Trial. JAMA Oncol. 2015 Oct;1(7):931-41. doi: 10.1001/jamaoncol.2015.2666. PMID 26247543
- [Background] Bekelman JE, Sylwestrzak G, Barron J, Liu J, Epstein AJ, Freedman G, Malin J, Emanuel EJ. Uptake and costs of hypofractionated vs conventional whole breast irradiation after breast conserving surgery in the United States, 2008-2013. JAMA. 2014 Dec 17;312(23):2542-50. doi: 10.1001/jama.2014.16616. PMID 25494006
- [Background] Jagsi R, Falchook AD, Hendrix LH, Curry H, Chen RC. Adoption of hypofractionated radiation therapy for breast cancer after publication of randomized trials. Int J Radiat Oncol Biol Phys. 2014 Dec 1;90(5):1001-9. doi: 10.1016/j.ijrobp.2014.09.032. PMID 25539365
- [Derived] Wong JS, Uno H, Tramontano AC, Fisher L, Pellegrini CV, Abel GA, Burstein HJ, Chun YS, King TA, Schrag D, Winer E, Bellon JR, Cheney MD, Hardenbergh P, Ho A, Horst KC, Kim JN, Leonard KL, Moran MS, Park CC, Recht A, Soto DE, Shiloh RY, Stinson SF, Snyder KM, Taghian AG, Warren LE, Wright JL, Punglia RS. Hypofractionated vs Conventionally Fractionated Postmastectomy Radiation After Implant-Based Reconstruction: A Randomized Clinical Trial. JAMA Oncol. 2024 Oct 1;10(10):1370-1378. doi: 10.1001/jamaoncol.2024.2652. PMID 39115975

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The following are reasons for withdrawal from the study before starting protocol treatment:
  * patients withdrew due to the treatment arm assignment
  * patients withdrew due to a change in treatment site
  * clinician withdrew patients due to tissue expander removal and other treatment needs
Groups:
- Arm 1: Hypofractionation: 16 fractions of radiation therapy (daily, Monday through Friday) to the chest wall with or without internal mammary nodes, and 15 fractions to the supraclavicular (with or without axillary) lymph nodes.
  Radiation Therapy: For the conventional fractionation arm: Each fraction will consist of 200 cGy per day. Total dose = 5000 cGy to the chest wall and 4600-5000 cGy to the lymph nodes.
  For the hypofractionation arm: Each fraction consists of 266 cGy per day. Total dose = 4256 cGy to the chest wall and 3990 cGy to the lymph nodes.
- Arm 2: Conventional Radiation Therapy: 25 fractions of radiation therapy (daily, Monday through Friday) to the chest wall with or without internal mammary nodes, and 23-25 fractions to the supraclavicular (with or without axillary) lymph nodes.
  Radiation Therapy: For the conventional fractionation arm: Each fraction will consist of 200 cGy per day. Total dose = 5000 cGy to the chest wall and 4600-5000 cGy to the lymph nodes.
  For the hypofractionation arm: Each fraction consists of 266 cGy per day. Total dose = 4256 cGy to the chest wall and 3990 cGy to the lymph nodes.
Period: Baseline
Arm/Group | Arm 1: Hypofractionation | Arm 2: Conventional Radiation Therapy
Started | 199 | 201
Completed | 192 | 199
Not Completed | 7 | 2
Not completed — Some participants skipped the survey question related to the primary outcome being analyzed. | 7 | 2
Period: 6-month Follow-up
Arm/Group | Arm 1: Hypofractionation | Arm 2: Conventional Radiation Therapy
Started | 192 | 199
Completed | 166 | 166
Not Completed | 26 | 33
Not completed — Withdrawal by subject, loss to follow-up | 26 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Hypofractionation | Arm 2: Conventional Radiation Therapy | Total
Number analyzed (Participants) | 199 | 201 | 400
Age, Customized [Count of Participants; unit: Participants]
  Age: <40 years | 42 | 41 | 83
  Age: 40-50 years | 84 | 90 | 174
  Age: 51-60 years | 49 | 42 | 91
  Age: 60+ years | 19 | 19 | 38
  Age: Missing | 5 | 9 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 201 | 400
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 27 | 46
  Not Hispanic or Latino | 180 | 174 | 354
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 12 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 157 | 161 | 318
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 20 | 35
Region of Enrollment [Number; unit: participants]
  United States | 199 | 201 | 400
Education [Count of Participants; unit: Participants]
  No College | 20 | 29 | 49
  Some college | 32 | 42 | 74
  College graduate | 63 | 57 | 120
  Some graduate/graduate degree | 80 | 72 | 152
  Missing | 4 | 1 | 5
BMI [Count of Participants; unit: Participants]
  <20 (kg/m^2) | 18 | 11 | 29
  20.0-24.9 (kg/m^2) | 79 | 75 | 154
  25.0-29.9 (kg/m^2) | 55 | 60 | 115
  30.0-34.9 (kg/m^2) | 30 | 34 | 64
  Greater than or equal to 35.0 (kg/m^2) | 16 | 20 | 36
  Missing | 1 | 1 | 2
Smoking Status [Count of Participants; unit: Participants]
  Never Smoked | 147 | 140 | 287
  Current/Former Smoker | 52 | 61 | 113
Prior Infection [Count of Participants; unit: Participants]
  No | 188 | 187 | 375
  Yes | 11 | 14 | 25
Cancer Laterality [Count of Participants; unit: Participants]
  Laterality: Right | 113 | 93 | 206
  Laterality: Left | 86 | 107 | 193
  Missing | 0 | 1 | 1
Hormone Receptor Status [Count of Participants; unit: Participants] — A pathologist tests the surgical specimen for expression of hormone receptors, like estrogen or progesterone.
  Participants
    Positive | 162 | 174 | 336
    Negative | 37 | 27 | 64
HER2 Status [Count of Participants; unit: Participants] — HER2 is a gene. To determine the HER2 status of breast cancer, a tumor sample is tested for either the number of copies of the HER2 gene, or for the amount of HER2 protein.
  Participants
    Equivocal | 11 | 11 | 22
    Negative | 146 | 149 | 295
    Positive | 42 | 39 | 81
    Unknown | 0 | 2 | 2
Histology [Count of Participants; unit: Participants]
  Invasive Ductal | 139 | 147 | 286
  Invasive Lobular | 29 | 32 | 61
  Both | 25 | 14 | 39
  Other | 6 | 8 | 14
Tumor Grade [Count of Participants; unit: Participants] — A pathologist looks at tumor samples under a microscope to see how much the cancer cells look like normal cells. If a tumor sample gets a low grade, those cells look more like normal breast cells. If a tumor sample gets a high grade, those cells look very different than normal breast cells.
  Participants
    Poorly Differentiated (Grade 3) | 82 | 78 | 160
    Moderately Differentiated (Grade 2) | 95 | 96 | 191
    Well Differentiated (Grade 1) | 20 | 26 | 46
    Not applicable | 2 | 1 | 3
Tumor Size [Count of Participants; unit: Participants]
  Less than or equal to 2 cm | 99 | 114 | 213
  Greater than 2 cm - Less than or equal to 5 cm | 60 | 49 | 109
  Greater than 5cm | 21 | 23 | 44
  Missing | 19 | 15 | 34
Lymphatic Vessel Invasion (LVI) [Count of Participants; unit: Participants]
  Negative | 118 | 126 | 244
  Other | 79 | 73 | 152
  Missing | 2 | 2 | 4
Total number of positive nodes [Count of Participants; unit: Participants]
  0 nodes | 56 | 52 | 108
  1 node | 65 | 76 | 141
  2 nodes | 33 | 32 | 65
  3 or more nodes | 38 | 34 | 72
  Missing | 7 | 7 | 14
Axillary Node Dissection [Count of Participants; unit: Participants]
  No | 99 | 112 | 211
  Yes | 100 | 89 | 189
Axillary Nodes Removed [Median (Full Range); unit: Nodes] | 8.5 [0 to 36] | 9.0 [0 to 27] | 9 [0 to 36]
Location of Device [Count of Participants; unit: Participants] — In this study, participants underwent immediate reconstructive surgery with placement of either a tissue expander or permanent implant at the time of mastectomy. "Device" refers to either the tissue expander or permanent implant.
  Participants
    Pre-pectoral | 115 | 118 | 233
    Sub-pectoral | 84 | 79 | 163
    Not applicable/Unknown | 0 | 4 | 4
Device irradiated [Count of Participants; unit: Participants] — In this study, participants underwent immediate reconstructive surgery with placement of either a tissue expander or permanent implant at the time of mastectomy. "Device" refers to either the tissue expander or permanent implant.
  Participants
    Expander | 160 | 156 | 316
    Implant | 39 | 45 | 84
Neoadjuvant Chemotherapy [Count of Participants; unit: Participants]
  Yes | 137 | 134 | 271
  No | 62 | 67 | 129
  Unknown | 0 | 0 | 0
Neoadjuvant endocrine therapy [Count of Participants; unit: Participants]
  Yes | 46 | 39 | 85
  No | 152 | 162 | 314
  Unknown | 1 | 0 | 1
Radiation Therapy [Count of Participants; unit: Participants] — Population: Number analyzed differs from overall number due to participant withdrawals or participants found to be ineligible.
  Participants
    number analyzed (Participants) | 194 | 192 | 386
    Chest Wall and Nodes | 170 | 160 | 330
    Chest Wall alone | 19 | 23 | 42
    Missing due to study withdrawal | 5 | 9 | 14
Technique [Count of Participants; unit: Participants] — Population: Number analyzed differs from overall number due to participant withdrawals or participants found to be ineligible.
  Participants
    number analyzed (Participants) | 194 | 192 | 386
    IMRT | 82 | 78 | 160
    3D-Conformal | 109 | 112 | 221
    Missing | 3 | 2 | 5
Time from surgery to RT (months) (Median, Q1, Q3) [Median (Inter-Quartile Range); unit: Months] | 2.7 [1.8 to 5.3] | 2.4 [1.8 to 4.9] | 2.5 [1.8 to 5.1]

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Outcomes Using the FACT-B
Description: The primary outcome is the change at 6 months from baseline in patient-reported outcomes on the Physical Well Being (PWB) sub-domain of the Functional Assessment of Cancer Therapy-Breast (FACT-B) instrument. The FACT-B is a 37-item instrument designed to measure five domains of health-related quality of life in breast cancer patients. The higher the score, the better the quality of life.
  Score ranges:
  * The score range for the FACT-B total score is 0-148.
  * The score range for the PWB, social/family well-being (SWB), and functional well-being (FWB) subscales is 0-28.
  * The score range for the emotional well-being (EWB) subscale is 0-24.
  * The score range for the breast cancer subscale (BCS) is 0-40.
Time Frame: 6 months
Population: Some participants skipped the survey questions related to the primary outcome being analyzed. This is why there is a discrepancy between the number analyzed for each domain and the total number of participants in each arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Hypofractionation | Arm 2: Conventional Radiation Therapy
Number analyzed (Participants) | 199 | 201
score on a scale
  Baseline FACT-B: number analyzed (Participants) | 186 | 192
  Baseline FACT-B | 104.3 (14.5) | 102.4 (17.0)
  Baseline PWB: number analyzed (Participants) | 187 | 195
  Baseline PWB | 22.4 (5.0) | 22.5 (4.7)
  Baseline SWB: number analyzed (Participants) | 186 | 194
  Baseline SWB | 23.8 (4.1) | 23.0 (4.6)
  Baseline EWB: number analyzed (Participants) | 188 | 193
  Baseline EWB | 16.2 (2.8) | 15.8 (3.5)
  Baseline FWB: number analyzed (Participants) | 187 | 193
  Baseline FWB | 16.7 (4.4) | 16.3 (4.8)
  Baseline BCS: number analyzed (Participants) | 187 | 195
  Baseline BCS | 25.3 (4.6) | 24.9 (5.2)
  6-month FACT-B: number analyzed (Participants) | 161 | 168
  6-month FACT-B | 105.0 (15.0) | 103.5 (17.7)
  6-month PWB: number analyzed (Participants) | 162 | 169
  6-month PWB | 23.0 (4.1) | 22.4 (4.7)
  6-month SWB: number analyzed (Participants) | 162 | 168
  6-month SWB | 22.4 (4.9) | 22.2 (5.0)
  6-month EWB: number analyzed (Participants) | 163 | 169
  6-month EWB | 16.5 (3.2) | 16.1 (3.8)
  6-month FWB: number analyzed (Participants) | 163 | 169
  6-month FWB | 17.7 (4.3) | 17.3 (4.5)
  6-month BCS: number analyzed (Participants) | 161 | 169
  6-month BCS | 25.4 (4.7) | 25.4 (5.4)

2. Secondary Outcome: Oncologic and Clinical Outcomes Assessed Using Medical Record Abstractions.
Description: Clinical and oncologic outcomes (rare radiation side effects, recurrence, infections, additional surgeries) will be assessed over a period of 10 years through annual medical record abstractions.
Time Frame: 10 years
Reporting Status: Not Posted

3. Secondary Outcome: Cosmetic Outcomes Assessed Using Photographic Evaluations.
Description: Cosmetic outcomes (quality of reconstructive surgery throughout and after radiation therapy) will be assessed from baseline to 18 months by trained physicians using a standardized rating scale.
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected if they occurred any time between initiation of protocol treatment and 3-years after the initiation of protocol treatment. All AEs reported throughout the study period are presented below in the data tables. Sites were asked to only report events listed in the Adverse Event Reporting Description. Some AEs below never occurred during the study period. Additional AEs that did not fall into these categories were also collected and reported.
Description: Reportable AEs include:
  * Grade 1, 2, or 3 brachial plexopathy
  * Grade 3 chest wall pain
  * Grade 3 lymphedema
  * Grade 3, 4, or 5 myocardial infarction
  * Grade 1, 2, 3, 4, or 5 pneumonitis
  * Grade 3, 4, or 5 treatment related secondary malignancy
  * Grade 3, 4, or 5 wound infection
  * Unexpected grade 3 or 4 with a possible, probable, or definite attribution to radiation therapy
  * Grade 5 (death): all deaths
Arm/Group | Arm 1: Hypofractionation | Arm 2: Conventional Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 2/199 | 2/201
Serious Adverse Events (participants affected / at risk) | 37/199 | 29/201
Other Adverse Events (participants affected / at risk) | 4/199 | 2/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Hypofractionation (N=199) | Arm 2: Conventional Radiation Therapy (N=201)
Distant recurrence (General disorders) | 11 | 12
Local-regional recurrence (General disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Infection (Infections and infestations) | 22 | 14 — Breast or wound infection
Lymphedema (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Hypofractionation (N=199) | Arm 2: Conventional Radiation Therapy (N=201)
Dehisence (Skin and subcutaneous tissue disorders) | 3 | 1
Capsular Contracture (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT03422003/Prot_SAP_000.pdf